CLINICAL TRIAL: NCT03309059
Title: Comparison Between the Effect of Zinc Oxide and Non-irritant Barrier Film on the Prevention of Incontinence-Associated Dermatitis in Hospitalized Elderly in a Teaching Hospital
Brief Title: Comparison of Barrier Products in the Prevention of Incontinence-associated Dermatitis in Hospitalized Elderly
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other)
Responsible Party: Principal Investigator, Carla Lucia Goulart Constant Alcoforado, Assistant Professor, Department of Basic Nursing, Federal University of Minas Gerais
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: x2mmdd79
Record Dates: First submitted 2017-01-15; First posted 2017-10-13 (Actual); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Diaper Rash
Keywords: Nursing care; diaper rash; fecal incontinence; urinary incontinence
MeSH Terms: conditions — Diaper Rash; Fecal Incontinence; Urinary Incontinence | interventions — Hydrotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- water and soap (Placebo Comparator): Will be composed of elderly patients who present with fecal and / or urinary incontinence and who, therefore, need to implement measures to prevent the development of IAD with the use of soap and water in the area and subsequent diaper placement disposable. This type of procedure is standardized in the medical clinic wards of the hospital under study, and for this reason, it was defined as control.
  Interventions: Device: water and soap
- zinc oxide (Active Comparator): will be composed of elderly patients who present with fecal and / or urinary incontinence and who, therefore, need to implement measures to prevent the development of IAD with the use of soap and water sanitation and application of zinc oxide . The patient presenting with urinary and / or fecal eliminations will undergo such intervention and then the placement of the disposable diaper used by the hospital.
  Interventions: Device: zinc oxide
- Non-Irritant Barrier Film (Experimental): will be composed of the elderly patients who present fecal and / or urinary incontinence and that, therefore, it is necessary to implement measures to prevent the development of ICD with the use of soap and water hygiene and application of Non Irritant Barrier Film. The patient who presents with urinary and / or fecal eliminations will undergo this intervention and then the placement of the disposable diaper used by the hospital.
  Interventions: Device: Non-Irritant Barrier Film

INTERVENTIONS:
Device: water and soap — Use of soap and water in the area and subsequent diaper placement disposable.
  Arms: water and soap
Device: zinc oxide — Use of soap and water sanitation and application of zinc oxide.
  Arms: zinc oxide
Device: Non-Irritant Barrier Film — Use of soap and water hygiene and application of Non Irritant Barrier Film.
  Arms: Non-Irritant Barrier Film

SUMMARY:
In clinical practice, there are a large number of patients hospitalized with Incontinence-Associated Dermatitis. Studies are needed to determine the effectiveness of products available for disease prevention. It is believed that the use of the non-irritant barrier film is superior to the use of zinc oxide in the prevention of Incontinence-Associated Dermatitis. The objective of this study is to compare the effect of the use of zinc oxide ointment with the use of non-irritant barrier film in the prevention of diaper dermatitis in incontinent patients admitted to medical clinic units.

DETAILED DESCRIPTION:
Introduction Skin lesions associated with moisture are defined as inflammation and skin erosion arising from prolonged exposure to sources such as urine, feces, sweat, wound exudate, mucus and saliva. They are initially triggered by lesions of the corneal extract, induced by exposure to multiple factors such as hyperhydration, friction, temperature, chemical irritants, urine and feces.

Among these types of lesions there is Incontinence Associated Dermatitis (IAD) which is a common clinical manifestation in patients with urinary and / or fecal incontinence. It is a skin inflammation that occurs as a consequence of the contact of the perineal, perigenital, perianal and adjacent areas with the urine and feces, besides erosion of the epidermis and macerated appearance.

The prevalence of IAD was reported as responsible for 7% of skin lesions in incontinent patients in nursing homes, 50% of them with fecal incontinence and 42% in hospitalized incontinent adults.

That the hospitalized incontinent individual is exposed to extrinsic and intrinsic factors that increase the susceptibility to IAD. As intrinsic factors, age, level of consciousness, oxygenation, mobility and comorbidity are mentioned, while extrinsic factors are related to exposure to incontinence, humidity and friction, as well as the frequency and quality of hygiene. Elderly incontinents are particularly vulnerable to the development of IAD because they have fewer layers of corneal extract, and also show a gradual decline in the barrier function associated with collagen and elastin decrease, as well as a decrease in microcirculation.

Patients bedridden, dependent, without sphincter control make constant use of diapers. In this universe of patients, the elderly are hospitalized. They demand more health services, hospitalizations are more common and hospitalization time is higher.

There is a high prevalence of chronic-degenerative diseases that imposes a need for greater hospitalization and progressive loss of the autonomy of the elderly. In this context, when IAD affects them, it is necessary to consider that the skin presents a sequence of alterations resulting from the aging process, making it more susceptible to the appearance of infections, wounds that consequently require a longer time for the process of aging. Healing occurs.

Demonstrate that the topic is little discussed by health professionals who care for the elderly population, and nursing has provided assistance based on experience gained in childcare, not based on scientific evidence to address the problem in Adults and the elderly. Thus, this situation may not address the needs of the care that the skin of the elderly may require.

The use of the diaper has been reported as one of those responsible for the appearance of dermatological disorders and exacerbation of episodes of urinary incontinence and decrease in the quality of life of these individuals. However, have identified specific care for the prevention and treatment of the IAD problem. However, they have not been tested and directed to the elderly population.

The measures are considered to be rather complex but relevant. For prevention, it is necessary to avoid or minimize exposure to causal factors by combining specific skin care, such as correct and gentle cleansing of the area, application of ointment or paste to protect against moisture and skin maceration.

Cleaning the skin with soap and water are traditionally used, as it is a common and necessary procedure, both at home and in the hospital. The wash removes organic debris from the surface of the skin, including scaly cells, fat and microorganisms. Water participates in the elimination of waste through mechanical and chemical action. The soap has surfactants that favor cleaning since they reduce the surface tension of the water, considering that the water in the soap also eliminates the residues. However, the surfactants contained in the soap can cause contact dermatitis, besides removing the hydrolipidic mantle by drying effect and thus weakening the protective function of the skin.

In addition to proper sanitization, the application of zinc oxide, which is a protective agent that promotes an occlusive barrier, is indicated which is able to prevent the passage of liquid from the inside out of the stratum corneum and prevents undesirable results from contact with urine And feces. It is commonly used due to its accessibility, resistance and cost, however, although it is more accessible, its long-term use may impose more costs on institutions.

A non-irritating alcohol-free product called Non-Irritant Barrier Film (PBNI) has been on the market since the 1990s. It is a mixture based on hexamethyldisiloxane, isoctane, thermopolymer acylate and polyphenylmethylsiloxane which upon contact with air forms a transparent, fluid impermeable, non-tissue irritating and non-cytotoxic film. It acts as a protection between skin and fluids and ease of application and removal, skin visibility and reduction of the frequency of incontinence-associated dermatitis are advantages of using film.

Defend the need for studies that present strong evidence for the prevention and treatment of IAD. In this sense, it is considered necessary to determine the efficacy of the products available for the prevention of the Nursing Diagnosis (ED) of Impaired Skin Integrity related to the use of diapers.

Considering these considerations, and due to the scarce knowledge about the best skin care of elderly patients with fecal and / or urinary incontinence, hospitalized in medical clinics indicated in the prevention of IAD, the following questions are asked: the use of the disposable diaper associated with Zinc oxide paste is more effective when compared to the use of disposable diaper associated with Non-Irritant Barrier Film in the prevention of incontinence-associated dermatitis?

Hypothesis H0 = The use of the disposable diaper associated with the previous cleaning with soap and water and subsequent application of zinc oxide is equivalent to the use of the disposable diaper associated with previous cleaning with soap and water and subsequent application of the non-irritating barrier film in the prevention of IAD In elderly incontinent patients admitted to a medical clinic.

H alternative = The use of the disposable diaper associated with cleaning with soap and water and subsequent application of Non Irritant Barrier Film is more effective in the prevention of IAD in elderly patients admitted to a medical clinic.

goal General objective To evaluate the effect of using zinc oxide ointment compared to Non-Irritant Barrier Film in the prevention of diaper dermatitis in elderly patients with faecal and / or urinary incontinence admitted to a medical clinic.

Specific objectives Identify risk factors for the development of impaired skin integrity related to faecal and / or urinary incontinence as evidenced by diaper area dermatitis in the hospitalized elderly population.

Identify changes in the skin in the diaper region during the use of the diaper with the application of zinc oxide.

Identify skin changes in the area of the diaper during the use of the diaper with the application of Non-Irritant Barrier Film.

Compare the best intervention for the prevention of diaper area dermatitis, a sign of impaired skin integrity, considering the need of the elderly population.

Outcome It will be considered a primary outcome of this study: whole skin in the area of diaper use with the use of soap and water and zinc oxide ointment; Skin integrity in the area of diaper use with the use of soap and water and Non-Irritant Barrier Film.

Population and Sample The population of this study will be composed of all the elderly patients who are bedridden and who present with discontinuation of the sphincter, who use a disposable diaper and who meet the inclusion criteria.

The sampling scheme used for data collection will be simple random sampling, within each of the groups studied. Thus, each sample unit within the population has the same probability of being selected to be part of the sample. In this study, a patient could be selected once, configuring a simple random sample without replacement.

To determine the minimum sample size required to detect significant differences between different treatments it is necessary to define a priori the minimum difference for which the test will present a significant result, the value of the desired power in addition to the level of significance of the test and the deviation Characteristics to be compared for the study population. The significance used to calculate the sample size will be 0.05. Thus, a significant difference will be considered for results whose probability of significance of the test, p-value, is less than or equal to 5%.

For this research, sample sizes were initially calculated considering power values at levels of 0.80 (80%), 0.90 (90%) and 0.95 (95%). The sample size was calculated considering the values of the statistical significance of the test, minimum significant difference in terms of 1, 0.75, 0.50 and 0.25 standard deviations and test power as described above.

The study by Chimentão and Domansky (2012) was used to calculate the prevalence of IAD in elderly patients in the nursing home (7%).

With these results, it was decided by a number of patients that will be part of the study of 79 for each of the groups studied. With this sample size it will be possible to identify differences from 0.5 standard deviations, with a power of 80% and a significance of 0.05.

The sample and the random allocation will be performed, using statistical technique and using a specific computer program. The time when this will be done will be as close as possible to the time of the intervention. The secrecy of the allocation list will be maintained.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older, exhibit stifle incontinence, wear disposable diapers, and be at risk for Incontinence-Associated Dermatitis

Exclusion Criteria:

* Patients with allergic reaction to the products used in the study

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2016-05; Primary Completion 2017-11 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Skin integrity assessment | Through the use of data collection instrument the skin will be evaluated at the 13 day follow up.
  The skin of the perineal, perigenital, perianal and adjacent regions will be evaluated for the presence of Incontinence-Associated Dermatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Tania C Machado Chianca, Phd, Study Director — Federal University of Minas Gerais; Flavia F Ercole, Phd, Study Chair — Federal University of Minas Gerais
Locations (1):
- Risoleta Tolentino Neves Hospital, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gray M, Black JM, Baharestani MM, Bliss DZ, Colwell JC, Goldberg M, Kennedy-Evans KL, Logan S, Ratliff CR. Moisture-associated skin damage: overview and pathophysiology. J Wound Ostomy Continence Nurs. 2011 May-Jun;38(3):233-41. doi: 10.1097/WON.0b013e318215f798. PMID 21490547
- [Background] Fernandes JD, Machado MC, Oliveira ZN. [Clinical presentation and treatment of diaper dermatitis--part II]. An Bras Dermatol. 2009 Jan-Feb;84(1):47-54. doi: 10.1590/s0365-05962009000100007. Portuguese. PMID 19377759
- [Background] ROCHA, N.; SELORES, M. Dermatite das fraldas. Nascer e Crescer- Revista do Hospital de Crianças Maria Pia. 2004:3 206-14
- [Background] BLISS, D.Z; LOWRY, A; WHITEBIRD, R; SAVIK, K; FAN, Q; JUNG, H.J. Absorbent product use and incontinence associated dermatitis in community-living persons with fecal incontinence. Abstracts of the 38th Annual Meeting of the International Continence Society; October, 2008 In: DOMANSKY, R.C; BORGES, E.L. Manual para prevenção de lesões de pele. Recomendações baseadas em evidências. RJ: Editora Rubio, 2012. 270p.
- [Background] AQUINO, A.L.; CHIANCA, T.C.M., BRITO R.C.S. Integridade da pele prejudicada, evidenciada por dermatite da área das fraldas: revisão integrativa. Rev. Eletr. Enf. [Internet]. 2012 abr/jun;14(2):414-24.
- [Background] Newman DK, Fader M, Bliss DZ. Managing incontinence using technology, devices, and products: directions for research. Nurs Res. 2004 Nov-Dec;53(6 Suppl):S42-8. doi: 10.1097/00006199-200411006-00007. PMID 15586147